CLINICAL TRIAL: NCT05385744
Title: An International, Multicenter, Randomized, Double-Blind, Double-Masked Study of the Efficacy and Safety of BCD-132 (JSC BIOCAD, Russia) Using an Active Reference Drug (Teriflunomide) for the Treatment of Patients With Multiple Sclerosis
Acronym: MIRANTIBUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-132-4
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — teriflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-132 (Experimental): IV infusion every 24 weeks in combination with daily placebo tablets. The total duration of the blinded therapy is 100 weeks (a total of 5 treatment cycles with BCD-132 in combination with the daily placebo tablets)
  Interventions: Biological: BCD-132
- Teriflunomide, 14 mg orally (Active Comparator): Teriflunomide, 14 mg orally daily, in combination with intravenous placebo infusions. The total duration of the blinded therapy is 100 weeks (a total of 5 treatment cycles with intravenous placebo infusions in combination with daily teriflunomide tablets).
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Biological: BCD-132 — anti-CD20 monoclonal antibody
  Arms: BCD-132
Drug: Teriflunomide — Teriflunomide 14 mg
  Arms: Teriflunomide, 14 mg orally

SUMMARY:
Clinical study BCD-132-4/MIRANTIBUS is an international, multicenter, randomized, double-blind, double-masked study using an active reference drug (teriflunomide). The goal of the study is to evaluate the efficacy and safety of BCD-132 in the treatment of patients with relapsing multiple sclerosis.

DETAILED DESCRIPTION:
Clinical study No. BCD-132-4/MIRANTIBUS is an international, multicenter, randomized, double-blind, double-masked study using an active reference drug (teriflunomide). The goal of the study is to evaluate the efficacy and safety of BCD-132 in the treatment of patients with relapsing multiple sclerosis.

The study includes adults with relapsing-remitting multiple sclerosis (according to 2017 revision to the McDonald Diagnostic Criteria for Multiple Sclerosis) and EDSS disability score up to 5.5.

Some of the subjects in this study will be patients rolled over from ongoing phase II clinical study No. BCD-132-2; treatment group, individual product kit number (IPKN), stratification factors, order of procedures and timeframes for blinded therapy with a duration of up to 100 weeks will remain the same.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation in the study;
2. Male and female subjects, 18 to 60 years of age
3. Diagnosis of relapsing multiple sclerosis (according to 2017 revision to the McDonald Diagnostic Criteria for Multiple Sclerosis);
4. Documentary evidence that, at the time of signing the informed consent, the subject had:

   1. at least 1 relapse within the last calendar year (12 months), or
   2. 2 relapses within the last 2 years (24 months), or
   3. at least 1 T1 gadolinium-enhanced brain lesion on MRI and 1 relapse within 2 calendar years (24 months) prior to signing the informed consent;
5. The subject must be neurologically stable for 30 days prior to signing the informed consent
6. Total EDSS score 0 to 5.5 inclusive
7. Positive anti-Varicella Zoster IgG antibodies according to screening test results;
8. Absence of suicidal ideation and behavior confirmed at screening according to C-SSRS score within 1 month prior to signing the informed consent
9. Willingness of both female and male patients and their sexual partners of childbearing potential to use reliable contraception

Exclusion Criteria:

Primary progressive MS; Duration of multiple sclerosis for more than 10 years with EDSS ≤2.0 according to screening assessments; Other disorders (besides multiple sclerosis), which could affect the assessment of symptom severity for the primary disease A relapse during screening period ; Use of systemic corticosteroids for 30 days prior to signing the informed consent; Disorders, besides multiple sclerosis, requiring long-term systemic therapy with corticosteroids and/or immunosuppressants; Heart failure (NYHA functional class III/IV); encephalopathy, lactic acidosis, MELAS syndrome), neuromyelitis optica, sarcoidosis; Diagnosis of HIV, hepatitis B, hepatitis C, or syphilis ; Increased TTG levels at least two times the upper limit of normal on screening tests; Suicidal ideation and/or behavior History of severe depression Pregnancy, breastfeeding, or intention to become pregnant at any point throughout the study period; Prior use of anti-B cell therapies Intolerance, including hypersensitivity to any component of BCD-132/teriflunomide, premedication drugs, or conditions in which the above drugs are contraindicated in the Investigator's opinion; History of severe allergic or anaphylactic reactions to humanized and/or murine monoclonal antibodies; History of progressive multifocal leukoencephalopathy Known alcohol or drug addiction or signs of current alcohol/drug addiction Inability to follow the procedures specified in the Protocol, as assessed by the Investigator;

Contraindications to MRI and administration of gadolinium-based contrast agents:

Any current or prior malignancies, except for successfully treated basal cell carcinoma and cervical carcinoma in situ Vaccination within 6 weeks prior to signing the informed consent

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Annualized relapse rate | week 48
  Annualized relapse rate at 48 weeks after the randomization of the last patient in the study

SECONDARY OUTCOMES:
Proportion of patients with persistent progression | week 48
  Persistent progression is defined as an increase in the EDSS score from Visit 1 by at least 1.0 in patients with a score >0 and ≤5.5 at the first visit and by at least 1.5 in patients with a score of 0 at the first visit
Total number of T1 Gd+ lesions | week 48
  Total number of T1 Gd+ lesions (per scan) detected on brain MRI;
CUA | week 48
  Combined unique active lesions
Proportion of patients without contrast-enhancing lesions | week 48
  Proportion of patients without contrast-enhancing lesions
Number of new or enlarged T2 lesions | week 48
  Number of new or enlarged T2 lesions
Proportion of patients without new or enlarged T2 lesions | week 48
  Proportion of patients without new or enlarged T2 lesions
Changes in the neurologic deficit according to EDSS score | week 48
  Changes in the neurologic deficit according to Expanded Disability Status Scale
Annualized relapse rate | week 48
  Mean annualized relapse rate
Proportion of patients with adverse reactions | week 48
Proportion of patients with serious adverse reactions | week 48

CONTACTS AND LOCATIONS:
Locations (1):
- State Budgetary Healthcare Institution of the Moscow Region M.F. Vladimirsky Moscow Regional Research and Clinical Institute, Moscow, Russia